CLINICAL TRIAL: NCT02918396
Title: The Substrate and Intervention Mechanisms for Persistent Atrial Fibrillation (SIMPle AF) Trial
Brief Title: The Substrate and Intervention Mechanisms for Persistent Atrial Fibrillation Trial
Acronym: SIMPle-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low enrollment of participants meeting eligibility criteria
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00084915
Record Dates: First submitted 2016-09-13; First posted 2016-09-29 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Atrial Fibrosis; Late Gadolinium Enhancement Magnetic Resonance Imaging; Computational Modeling; Rotor Anchor Sites
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional PVI (Active Comparator): Conventional PVI by Radio-frequency Ablation: Wide area circumferential pulmonary vein isolation (PVI) only (current standard of care) using radio-frequency ablation catheters.
  Interventions: Device: Conventional PVI by Radio-frequency Ablation
- PVI + Scar-based ablation (Experimental): Scar-Based Radio-frequency Ablation: Pulmonary vein isolation followed by targeting, using radio-frequency ablation, of dense LGE sites on MRI, which are confirmed on bipolar mapping to have voltage <0.3 mV.
  Interventions: Device: Scar-Based Radio-frequency Ablation
- PVI + Modeling-predicted rotors ablation (Experimental): Rotor Anchors Radio-frequency Ablation: Pulmonary vein isolation followed by radio-frequency ablation of rotor anchors predicted by modeling.
  Interventions: Device: Rotor Anchors Radio-frequency Ablation

INTERVENTIONS:
Device: Scar-Based Radio-frequency Ablation — Left atrial (LA) myocardium will be manually segmented prior to the procedure and 3D-volumes of the atrial anatomy with superimposed dense LGE maps will be generated. Prior to the PVI, a dense voltage map of the left atrium will be performed (>1000 points) iin sinus rhythm. After PVI, low voltage areas (defined as <0.3 mV) which are superimposed on dense LGE on the MRI will be targeted by radio frequency ablation with a contact force sensing, irrigated radiofrequency catheter approved by FDA for the treatment of atrial fibrillation.
  Arms: PVI + Scar-based ablation
Device: Rotor Anchors Radio-frequency Ablation — Left atrial (LA) myocardium will be manually segmented prior to the procedure and the LA shell, along with the LGE-MRI will be sent to the biomedical engineering team who will generate a 3D-model of the LA along with rotor anchor sites predicted by modeling. After the PVI, the 3D models will be displayed and the rotor anchor sites will be targeted by radiofrequency ablation with a contact force sensing, irrigated radiofrequency catheter approved by FDA for the treatment of atrial fibrillation.
  Arms: PVI + Modeling-predicted rotors ablation
Device: Conventional PVI by Radio-frequency Ablation — Conventional wide area circumferential ablation (WACA) pulmonary vein isolation will be performed using a contact-force sensing, irrigated radiofrequency catheter approved by FDA for the treatment of atrial fibrillation.
  Arms: Conventional PVI

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia with increasing morbidity and mortality. A catheter-based AF ablation technique that isolates pulmonary veins (PV) from the left atrium has been established to disrupt AF. Despite significant development, AF ablation with pulmonary vein isolation (PVI) is reported to have a success rate of 40-80% in various AF populations.

Persistent AF appears to be more reliant upon fibroblast proliferation and myocyte-fibroblast coupling than paroxysmal AF with obvious implications on its management. Despite the knowledge that fibrotic substrate is responsible for the perpetuation of persistent AF, several ablation techniques targeting these extra-pulmonary veins sites have failed to prove an additional benefit to PVI alone. Nevertheless, two recently developed technologies, aimed at detecting AF substrate with high precision, seem to constitute a potential breakthrough in the management of persistent AF. On one hand, late gadolinium-enhanced MRI (LGE-MRI) is a well-established method to identify fibrosis in the myocardium. Recent reports from a single center have shown that MRI-based left atrial fibrosis detection is able to predict the outcome of the procedure. Hence, targeting lesions seen on LGE-MRI in the setting of persistent AF is an option yet to be explored and compared to the widely adopted, yet suboptimal, PVI. On another hand, a novel ablation method with promising results is focal impulse and rotor modulation (FIRM). Undergoing wide sampling of the atria with spatiotemporal and computational mapping while in AF has identified areas with stable organized rotational electrical activity (rotors). Several studies are under way to prove the reproducibility of rotor mapping, with more groups reporting improved rates of acute and long-term suppression of AF with ablation of FIRM-identified rotors.

The SIMPle AF study will be a randomized clinical trial designed to test the hypothesis that ablation tailored to the underlying substrate using either LGE-detected dense scar or rotor anchor sites predicted by computational modeling is superior to anatomic non-tailored PVI ablation in patients with persistent AF. For the present study, the investigators plan to enroll a total of 30 patients.

DETAILED DESCRIPTION:
Objectives The main objective of the study is to identify the optimal ablation strategy for suppression of persistent AF.

The secondary objectives of the study are:

* To define the local myocardial image characteristics of slow conduction AF substrates.
* To define the local myocardial structural changes post ablation that associate with AF suppression at 1-year follow-up
* To compare cardiac remodeling and atrial function at 1-year follow-up between PVI only and tailored catheter ablation groups

Background

Atrial fibrillation (AF) is associated with increased risk for mortality, heart failure, and thromboembolic events, and has a worldwide prevalence of >33.5 million. Catheter ablation of AF is evolving as an effective therapy for symptomatic AF. Recurrent AF after ablation, however, remains a problem and has been reported to associate with the baseline extent of left atrial (LA) late gadolinium enhancement (LGE) on cardiac magnetic resonance (CMR). Mechanistically, persistent AF appears to be more reliant upon fibroblast proliferation and myocyte-fibroblast coupling than paroxysmal AF, which is primarily dependent upon pulmonary vein triggers. Therefore, the investigators hypothesize that the substrate for persistent AF is detectable on atrial LGE-CMR and variable among patients, and that the substrate predicts patient outcomes after anatomic non-tailored ablation, and is more likely to respond to individually tailored ablation approaches. Two individually tailored approaches will be studied including empiric targeting of dense LGE, confirmed on bipolar mapping to have voltage <0.3 mV, and modeling based targeting of rotor anchor sites.

Study Design

Initially, the investigators propose prospective enrollment of 30 participants with persistent AF. Patients presenting to the institution who meet the inclusion criteria will be asked to participate in the study. All patients will undergo routine clinical care including echocardiography as indicated.

All patients will undergo a LGE-MRI within 30 days prior to the ablation procedure. The clinical purpose of the initial MRI is to define the anatomy of the heart chambers as well as the vessels for procedure planning. For research purposes, the investigators will use this initial clinical MRI to delineate atrial structural remodeling or fibrosis to be used during the procedure in patients randomized to group 2 (pulmonary vein isolation + scar-based ablation) and for later analysis in all patients.

Imaging is done at the institution and will be reviewed for quality by the study staff. LGE-MRI sequences that do not meet quality standards for fibrosis analysis will not be further processed and these patients will be excluded from the study. Subjects for whom images are successfully evaluated will be randomized to the study groups.

This will be followed by block randomization in 1:1:1 format to a) pulmonary vein isolation (PVI) only (current standard of care), b) PVI plus targeting of dense LGE sites, which are confirmed on bipolar mapping to have voltage <0.3 mV, and c) PVI plus targeting of rotor anchor sites predicted by modeling.

At baseline, all patients will be evaluated for their quality of life (QOL) using the Short-form health survey (SF-36) for overall as well as AF-related impact on quality of life. The severity of symptoms will also be tested using the European Heart Rhythm Association (EHRA) score of atrial fibrillation. Clinical data will be stored electronically and linked to a specific research number. Information linking de-identified data to the patients will be stored in the locked research office, in a password-protected file. Only members of the research team, in charge of collecting clinical information, will have access to this file. Individual subject binders containing signed consent forms and clinical source documentation will be labeled using study subject numbers and stored in the locked research office mentioned previously.

A pre-ablation cardiac MRI is clinically indicated to assess baseline cardiac anatomy prior to procedure. Routine and LGE protocols will be used to acquire MR images. All patients will be asked to undergo a repeat LGE-MRI 12 months after the ablation. This is done for research purposes. Renal function is routinely monitored prior to gadolinium-enhanced MRI as a standard of clinical care.

With regards to the ablation procedure, all patients will undergo AF ablation. The procedure consists of circumferential pulmonary vein lesions under electro-anatomical guidance using CARTO (Biosense Webster Inc., Diamond Bar, CA). Operators will use either a 3.5mm irrigated tip radiofrequency ablation catheter (ThermoCool Smart-Touch, Biosense Webster Inc., Diamond Bar, CA) or a cryoballoon catheter (Arctic Front Advance, Medtronic Inc., Minneapolis, MN). This procedure is FDA approved and will be conducted in all treatment arms according to standard of care. However, patients in the second group will undergo additional targeting of dense LGE sites, confirmed on bipolar mapping to have voltage <0.3 mV and patients in the third group will undergo targeting of rotor anchor sites as predicted by computational modeling. A detailed protocol of rotor ablation is described in the literature and shows no added complications compared to the conventional procedure.

To prevent short-term recurrence of AF, patients will be kept on anti-arrhythmic regimen for the first 1 to 3 months after the ablation to be discontinued thereafter in the absence of AF recurrence, at the discretion of the treating physician. In addition, standard protocols for anticoagulation prior to, during, and after the ablation procedure will be applied.

After the ablation, clinical follow-up visits are scheduled at 3, 6 and 12 months. Research follow-up questionnaires and 12-lead ECG recordings will be done at the same day of the visits. All patients will undergo rhythm monitoring to detect AF recurrence using a portable, smart phone operated, AliveCor® Mobile ECG device.This device will be provided to the patients at no cost after enrollment in the study.

After the procedure, follow-up will be done on a weekly basis through trans-telephonic transmissions of ECG recordings. Periodic reminders will be sent to patients (via telephone, email, or mail) regarding follow up transmissions in the event that a weekly transmission is missed. In addition, study participants will be advised to provide recordings if they experience heart-related symptoms (palpitations, shortness of breath, rapid heartbeat, chest pain). This extensive rhythm monitoring protocol is not standard of care and is done for research purposes. Review of the rhythm monitoring data will be performed in accordance with current clinical guidelines. The device software and the investigators will analyze rhythm strips and a report will be available to the research team and to the treating physician upon his/her request. In addition, upon detection of any arrhythmia with important clinical implications, the investigators will notify the electrophysiologist involved in the care of the patient. The research team may contact the patient directly if prompt action is advised, such as reporting to the local emergency room or following up with their electrophysiologist. The rhythm monitoring protocol utilized in this study may result in unscheduled visits to the physician. If a repeat ablation procedure is indicated, it will be scheduled according to standards of clinical care.

Study duration and visits.

The investigators aim to complete the proposed study protocol in two years. After the ablation, patients will be followed at 3, 6 and 12 months via in clinic visit; a 1 month and 9 month follow up will take place via remote ECG transmission. Follow-up research questionnaires and post-ablation MRI will be scheduled to coincide with the routine clinical visits. Hence, no additional visits will be required of research participants unless it was not possible to schedule the MRI on the same day as clinic visits. Only then will the investigators ask participants to present to the institution for the follow-up MRI.

Study Statistics

Based on the variable success rate of 40-80% in AF ablation, the investigators anticipate that the study cohort of 30 patients would produce adequate sample size in all treatment arms and be sufficient to make meaningful statistical comparison.

Comparison variables will be presented as means +/- standard deviation, and categorical variables as numbers and percentages. Differences between treatment groups will be assessed using the Pearson Chi-square test and the Wilcoxon rank-sum test. Survival curves for time to event analysis will be estimated using the Kaplan-Meier method, and the differences between the curves will be tested for significance with the log-rank statistic. Weekly event rates will be calculated by dividing the event rate by the maximum follow-up period in each arm of the Kaplan-Meier analysis. Hazard ratios will be calculated by univariate and multivariate analysis using the Cox proportional-hazards regression model. When comparing MR image characteristics as well as LA function between pre and post-ablation imaging, the Student's t-test will be using for comparison of the means. All statistical testing will be 2-tailed. Results will be considered statistically significant at a level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* History of persistent atrial fibrillation
* Indicated for an AF-ablation procedure
* Agree to participate in the trial

Exclusion Criteria:

* Are unable or unwilling to provide informed consent for the SIMPle AF study
* Patients with cardiac devices like pacemakers, internal cardiac defibrillators and Cardiac Resynchronization Therapy Device (CRT). Patients with acute or chronic renal insufficiency (glomerular filtration rate <30 ml/min/1.73 m2), or patients in the perioperative liver transplantation period
* Pregnant women
* Patients who are unable to adhere to the follow up protocol
* Patients with contraindication to MRI, including ferromagnetic aneurysm clips, metal in the eye, and implanted ferromagnetic or other MRI-incompatible devices
* Patients in whom the LGE Cardiac MRI does not meet quality standards for fibrosis analysis
* Subjects without daily access to a smart phone or tablet compatible with the mobile-based application and ability to upload ECG tracings for the follow up period
* Patients with a history of allergic reactions to gadolinium-based contrast agents or ingredients and will not be premedicated**

  * Subjects with a history of reaction to contrast may be premedicated according to institutional protocol prior to receiving intravenous contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saman Nazarian, MD, PhD, Principal Investigator — Hospital of the University of Pennsylvania; Johns Hopkins Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akoum N, Marrouche N. Assessment and impact of cardiac fibrosis on atrial fibrillation. Curr Cardiol Rep. 2014 Aug;16(8):518. doi: 10.1007/s11886-014-0518-z. PMID 24950676
- [Background] Akoum N, Morris A, Perry D, Cates J, Burgon N, Kholmovski E, MacLeod R, Marrouche N. Substrate Modification Is a Better Predictor of Catheter Ablation Success in Atrial Fibrillation Than Pulmonary Vein Isolation: An LGE-MRI Study. Clin Med Insights Cardiol. 2015 Apr 27;9:25-31. doi: 10.4137/CMC.S22100. eCollection 2015. PMID 25983561
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D. 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design. Europace. 2012 Apr;14(4):528-606. doi: 10.1093/europace/eus027. Epub 2012 Mar 1. No abstract available. PMID 22389422
- [Background] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Background] Dorian P, Cvitkovic SS, Kerr CR, Crystal E, Gillis AM, Guerra PG, Mitchell LB, Roy D, Skanes AC, Wyse DG. A novel, simple scale for assessing the symptom severity of atrial fibrillation at the bedside: the CCS-SAF scale. Can J Cardiol. 2006 Apr;22(5):383-6. doi: 10.1016/s0828-282x(06)70922-9. PMID 16639472
- [Background] Estes NA 3rd, Sacco RL, Al-Khatib SM, Ellinor PT, Bezanson J, Alonso A, Antzelevitch C, Brockman RG, Chen PS, Chugh SS, Curtis AB, DiMarco JP, Ellenbogen KA, Epstein AE, Ezekowitz MD, Fayad P, Gage BF, Go AS, Hlatky MA, Hylek EM, Jerosch-Herold M, Konstam MA, Lee R, Packer DL, Po SS, Prystowsky EN, Redline S, Rosenberg Y, Van Wagoner DR, Wood KA, Yue L, Benjamin EJ. American Heart Association atrial fibrillation research summit: a conference report from the American Heart Association. Circulation. 2011 Jul 19;124(3):363-72. doi: 10.1161/CIR.0b013e318224b037. Epub 2011 Jun 27. No abstract available. PMID 21709057
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Inoue K, Kurotobi T, Kimura R, Toyoshima Y, Itoh N, Masuda M, Higuchi Y, Date M, Koyama Y, Okamura A, Iwakura K, Fujii K. Trigger-based mechanism of the persistence of atrial fibrillation and its impact on the efficacy of catheter ablation. Circ Arrhythm Electrophysiol. 2012 Apr;5(2):295-301. doi: 10.1161/CIRCEP.111.964080. Epub 2011 Oct 31. PMID 22042883
- [Background] Marrouche NF, Wilber D, Hindricks G, Jais P, Akoum N, Marchlinski F, Kholmovski E, Burgon N, Hu N, Mont L, Deneke T, Duytschaever M, Neumann T, Mansour M, Mahnkopf C, Herweg B, Daoud E, Wissner E, Bansmann P, Brachmann J. Association of atrial tissue fibrosis identified by delayed enhancement MRI and atrial fibrillation catheter ablation: the DECAAF study. JAMA. 2014 Feb 5;311(5):498-506. doi: 10.1001/jama.2014.3. PMID 24496537
- [Background] McGann C, Akoum N, Patel A, Kholmovski E, Revelo P, Damal K, Wilson B, Cates J, Harrison A, Ranjan R, Burgon NS, Greene T, Kim D, Dibella EV, Parker D, Macleod RS, Marrouche NF. Atrial fibrillation ablation outcome is predicted by left atrial remodeling on MRI. Circ Arrhythm Electrophysiol. 2014 Feb;7(1):23-30. doi: 10.1161/CIRCEP.113.000689. Epub 2013 Dec 20. PMID 24363354
- [Background] Narayan SM, Baykaner T, Clopton P, Schricker A, Lalani GG, Krummen DE, Shivkumar K, Miller JM. Ablation of rotor and focal sources reduces late recurrence of atrial fibrillation compared with trigger ablation alone: extended follow-up of the CONFIRM trial (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation). J Am Coll Cardiol. 2014 May 6;63(17):1761-8. doi: 10.1016/j.jacc.2014.02.543. Epub 2014 Mar 13. PMID 24632280
- [Background] Narayan SM, Krummen DE, Shivkumar K, Clopton P, Rappel WJ, Miller JM. Treatment of atrial fibrillation by the ablation of localized sources: CONFIRM (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation) trial. J Am Coll Cardiol. 2012 Aug 14;60(7):628-36. doi: 10.1016/j.jacc.2012.05.022. Epub 2012 Jul 18. PMID 22818076
- [Background] Runge VM. Safety of magnetic resonance contrast media. Top Magn Reson Imaging. 2001 Aug;12(4):309-14. doi: 10.1097/00002142-200108000-00007. PMID 11687717
- [Background] Schenck JF. Safety of strong, static magnetic fields. J Magn Reson Imaging. 2000 Jul;12(1):2-19. doi: 10.1002/1522-2586(200007)12:13.0.co;2-v. PMID 10931560
- [Background] Schnabel RB, Yin X, Gona P, Larson MG, Beiser AS, McManus DD, Newton-Cheh C, Lubitz SA, Magnani JW, Ellinor PT, Seshadri S, Wolf PA, Vasan RS, Benjamin EJ, Levy D. 50 year trends in atrial fibrillation prevalence, incidence, risk factors, and mortality in the Framingham Heart Study: a cohort study. Lancet. 2015 Jul 11;386(9989):154-62. doi: 10.1016/S0140-6736(14)61774-8. Epub 2015 May 7. PMID 25960110
- [Background] Shivkumar K, Ellenbogen KA, Hummel JD, Miller JM, Steinberg JS. Acute termination of human atrial fibrillation by identification and catheter ablation of localized rotors and sources: first multicenter experience of focal impulse and rotor modulation (FIRM) ablation. J Cardiovasc Electrophysiol. 2012 Dec;23(12):1277-85. doi: 10.1111/jce.12000. Epub 2012 Nov 6. PMID 23130890
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035
- [Background] Wilber DJ. Fibroblasts, focal triggers, and persistent atrial fibrillation: is there a connection? Circ Arrhythm Electrophysiol. 2012 Apr;5(2):249-51. doi: 10.1161/CIRCEP.111.968750. No abstract available. PMID 22511658
- [Background] Zareian M, Ciuffo L, Habibi M, Opdahl A, Chamera EH, Wu CO, Bluemke DA, Lima JA, Venkatesh BA. Left atrial structure and functional quantitation using cardiovascular magnetic resonance and multimodality tissue tracking: validation and reproducibility assessment. J Cardiovasc Magn Reson. 2015 Jul 1;17(1):52. doi: 10.1186/s12968-015-0152-y. PMID 26126732

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional PVI | PVI + Scar-based Ablation | PVI + Modeling-predicted Rotors Ablation
Started | 2 | 1 | 2
Completed | 2 | 1 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional PVI | PVI + Scar-based Ablation | PVI + Modeling-predicted Rotors Ablation | Total
Number analyzed (Participants) | 2 | 1 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 62 [58 to 66] | 74 [74 to 74] | 65 [60 to 70] | 65.6 [58 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 2 | 0 | 2 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 2 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of Atrial Fibrillation (AF) > 30 Seconds
Description: Primary outcome is defined as symptomatic or asymptomatic AF of at least 30 seconds duration that is documented by an ECG or mobile rhythm monitoring device (AliveCor), occurring after the 3-month blanking period following catheter ablation and up to 12 months.
Time Frame: Following the 90 day blanking period up to 12 months post-index pulmonary vein isolation
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional PVI | PVI + Scar-based Ablation | PVI + Modeling-predicted Rotors Ablation
Number analyzed (Participants) | 2 | 1 | 2
Participants | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | Conventional PVI | PVI + Scar-based Ablation | PVI + Modeling-predicted Rotors Ablation
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT02918396/Prot_SAP_000.pdf